CLINICAL TRIAL: NCT03710863
Title: Phase 2 Study of Intermittent Oral Dosing of CM082 in Patients With wAMD: Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy
Brief Title: Safety and Tolerability of Oral CM082 in Patients With wAMD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Collaborators: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-OPH-102
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — vorolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 Tablet (Experimental): Code Name: CM082 Tablet Other Name: X-82 Dosage and Administration: 25/50mg BID, P.O., two-week on/two-week off in four-week cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CM082

INTERVENTIONS:
Drug: CM082 — Subjects will receive CM082 orally twice daily for two weeks followed by two weeks off in four-week cycles. The starting dose of 25mg BID will be increased by 100% to the maximum dose of 50mg BID.The treatment period is tentatively set at 1 year.
  Other Names: X-82

SUMMARY:
This is a Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Intermittent Oral Dosing of CM082 tablets in Chinese Patients With wAMD.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase II Study to Evaluate the safety, tolerability, pharmacokinetics and preliminary Efficacy of intermittent oral dosing of CM082 tablets in Chinese patients with wAMD. The study will be performed in two different parts, dose-escalation phase (Part 1) and dose-expansion phase (Part 2). Subjects will receive CM082 orally twice daily for two weeks followed by two weeks off in four-week cycles. There are two dose levels, 25mg BID and 50mg BID. In part 1, the starting dose of 25mg BID(n=8) will be increased by 100% to the maximum dose of 50mg BID(n=8) if the number of patients who experience dose-limiting toxicities is less than 2 during the first cycle. In part 2, based on the relevant data from the dose escalation study, an expanded enrollment study was conducted at a safe and effective dose.Per dose group will enroll 12-24 patients. All patients will take CM082 until disease progression or unacceptable toxicity. The assessment of the safety and efficacy will be done every four weeks from 2nd-6th cycle and every 12 weeks after. Also, single/multiple dose pharmacokinetics in these patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization (CNV) associated with AMD, as evidenced on fluorescein angiography (FA) and OCT.
* Patients with either no previous anti-VEGF therapy or prior anti-VEGF therapy with the discontinuation time is at least 5 drug half-lives.
* ETDRS BCVA 20/400 to 20/32 in the study eye(s).
* Adequate bone marrow, hepatic, and renal functions.
* Willing to sign the ICF and comply with the study protocol.

Exclusion Criteria:

* Patients with Polypoidal Choroidal Vasculopathy (PCV) as evidenced on Indocyanine Green Angiography (ICG).
* Geographic atrophy involving the foveal center in the study eye.
* Previous treatment with photodynamic therapy (PDT), external beam radiation, subfoveal focal laser photocoagulation, submacular surgery or transpupillary thermotherapy.
* CNV due to causes other than AMD, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia.
* Any significant disease in the study eye that could compromise best-corrected visual acuity.
* Clinically significant impaired renal or hepatic function.
* Stroke within 12 months of the first dose or transient ischemic attack within 12 months of the first dose.
* Symptomatic congestive heart failure, unstable angina, acute coronary syndrome, myocardial infarction or coronary artery revascularization, or arterial thrombosis within 6 months of start of study drug, inadequately controlled hypertension, or ventricular tachyarrhythmias requiring ongoing treatment.
* QTc≥450 msec or subjects with a history of risk factors for Torsades de Pointes or other severe ECG abnormalities which are clinically relevant.
* Trabeculectomy or aqueous shunt or valve in the study eye.
* Use of any investigational agent or participation in any other clinical trial of an investigational agent or investigational therapy within thirty (30) days of the first dose.
* Allergy to the ingredients of the study drug.
* Women of childbearing age who are pregnant, breast-feeding or not using medically acceptable contraception; males who are unwilling to take adequate contraceptive measures.
* Need to take any medicine that is a strong inhibitor or inducer of CYP3A4.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | the first cycle(the first four weeks)
  Any serious adverse event in eye or any ≥3 grade adverse reactions cannot be reduced to below grade 3 after treatment for more than 7 days.

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | 8 weeks
  Change from baseline in mean BCVA (ETDRS)
Change in Choroidal Neovascularization (CNV) size | 8 weeks
  Change from baseline in mean CNV size (OCTA, FA/ICG)
Change in Central Retinal Thickness | 8 weeks
  Change from baseline in mean central retinal thickness (OCT)
Change in ERG | 8 weeks
  Change from baseline in ERG
Proportion Who Develop CNV in the Unaffected Fellow Eye | 8 weeks
  Diagnosis by FA

CONTACTS AND LOCATIONS:
Overall Officials: Yin Shen, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Hubei General Hospital, Wuhan, Hubei, China